CLINICAL TRIAL: NCT06917157
Title: Latency Antibiotics for Previable Rupture Of Membranes: LAPROM Trial
Brief Title: Latency Antibiotics for Previable Rupture Of Membranes Trial
Acronym: LAPROM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Khalil Chahine, House Staff, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-1285
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Preterm Prelabor Rupture of Membranes (PPROM)
Keywords: prophylactic antibiotics; neonatal morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of antibiotics prophylactically at the time of membrane rupture (Experimental): Membrane rupture per inclusion criteria will be less than 22 weeks
  Interventions: Drug: Administration of antibiotics prophylactically at the time of membrane rupture
- Administration of antibiotics non-prophylactically at 22 weeks (Active Comparator)
  Interventions: Drug: Administration of antibiotics non-prophylactically at 22 weeks

INTERVENTIONS:
Drug: Administration of antibiotics prophylactically at the time of membrane rupture — Participants will receive the antibiotic regimen:
  * Day 1: Oral Azithromycin 1 g once and intravenous Ampicillin 2 g every 6 hours
  * Day 2: Intravenous Ampicillin 2 g every 6 hours
  * Days 3-7: Oral Amoxicillin 500 mg every 8 hours
  Arms: Administration of antibiotics prophylactically at the time of membrane rupture
Drug: Administration of antibiotics non-prophylactically at 22 weeks — Participants will receive latency antibiotics starting 22 weeks 0 days:
  * Day 1: Oral Azithromycin 1 g once and intravenous Ampicillin 2 g every 6 hours
  * Day 2: Intravenous Ampicillin 2 g every 6 hours
  * Days 3-7: Oral Amoxicillin 500 mg every 8 hours
  Arms: Administration of antibiotics non-prophylactically at 22 weeks

SUMMARY:
The purpose of this study is to see if the use of prophylactic antibiotics in the expectant management of PPROM less than 22 weeks significantly reduce the rate of delivery within 7 days and to see if the use of prophylactic antibiotics in the expectant management of PPROM between 20 and 22 weeks decrease composite neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Preterm premature rupture of membranes at less than 22 weeks.
* Membrane rupture had occurred within 36 hours of randomization.
* Cervical dilatation is 3 cm or less (on visual or clinical examination).
* 4 or fewer contractions in the 60-minute monitoring period before randomization.
* Singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age
* Gestational age at randomization less than 22 weeks (≤21 weeks and 6 days) based on clinical information.

Exclusion Criteria:

* Nonreasoning fetal testing
* Vaginal bleeding
* Maternal or fetal indication for immediate delivery
* Cervical cerclage in place
* Receipt of latency antibiotics prior to randomization (azithromycin, ampicillin, or amoxicillin)
* Allergy to Penicillins or Azithromycin
* Febrile illness requiring antibiotics
* Placenta previa
* Multifetal gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that delivered their babies after membrane rupture | from baseline to day 7

SECONDARY OUTCOMES:
Latency, defined as the duration between rupture of membranes and delivery | from rupture of membranes to delivery(about 1-126 days after baseline)
Number of participants that have Chorioamnionitis | Baseline upto delivery (about 1-126 days after baseline)
Number of participants that develop sepsis | From baseline upto discharge (about 1-4 days post delivery)
Number of maternal deaths | From baseline upto discharge (about 1-4 days post delivery)
Number of admissions to intensive care unit (ICU) | From baseline upto discharge (about 1-4 days post delivery)
Number of participants that develop postpartum hemorrhage | From baseline upto discharge (about 1-4 days post delivery)
  postpartum hemorrhage could occur during the following:
  1. Transfusion
  2. Non-elective hysterectomy
  3. Use of two or more uterotonics other than oxytocin
  4. Other surgical interventions such as uterine compression sutures, uterine artery ligation, embolization and hypogastric ligation, balloon tamponade
  5. Curettage
Number of participants that develop maternal postpartum infection | within 6 weeks of delivery
  Infection is defined as one of the following:
  * Clinical diagnosis of endometritis
  * Wound reopened for hematoma, seroma, infection or other reasons
  * Cellulitis requiring antibiotics
  * Pneumonia
  * Pyelonephritis
  * Bacteremia unknown source
  * Septic pelvic thrombosis
Number of participants that develop maternal venous thromboembolism | within 6 weeks of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Chahine, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No